CLINICAL TRIAL: NCT06166121
Title: A Randomized, Double-blind, Placebo-controlled Study of ShenJu in the Treatment of Hyperlipidemia Combined With Carotid Atherosclerosis
Brief Title: Study on Hyperlipidemia Combined With Carotid Atherosclerosis With ShenJu Granules
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangdong Provincial Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Lei Wang,MD, Chief Physician, Guangdong Provincial Hospital of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: YF2022-215
Record Dates: First submitted 2023-05-06; First posted 2023-12-12 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Hyperlipidemia; Carotid Atherosclerosis
Keywords: Hyperlipidemia; Carotid arteriosclerosis; baPWV
MeSH Terms: conditions — Hyperlipidemias; Carotid Artery Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ShenJu (Experimental): On the basis of standardized drug treatment for Hyperlipidemia combined with carotid atherosclerosis, participants who met the inclusion criteria were randomly given ShenJu intervention on the day of inclusion, taking it twice a day for 90 days.
  Interventions: Other: ShenJu
- placebo (Placebo Comparator): On the basis of standardized drug treatment for Hyperlipidemia combined with carotid atherosclerosis, participants who met the inclusion criteria were randomly given placebo granules on the day of inclusion, which were taken twice a day for 90 days (the placebo was basically the same as ShenJu in terms of appearance, shape, color, taste, etc.)
  Interventions: Other: Placebo

INTERVENTIONS:
Other: ShenJu — One package per time, twice a day, 90 days of treatment
  Arms: ShenJu
Other: Placebo — One package per time, twice a day, 90 days of treatment (the placebo was basically the same as ShenJu in terms of appearance, shape, color, taste, etc.)
  Arms: placebo

SUMMARY:
This study focuses on PWV as the main outcome, aiming to evaluate the efficacy and safety of ShenJu in treating patients with hyperlipidemia combined with carotid atherosclerosis, and provide a basis for traditional Chinese medicine treatment of hyperlipidemia combined with carotid atherosclerosis.

DETAILED DESCRIPTION:
Hyperlipidemia is very harmful and easy to cause atherosclerosis. Atherosclerosis is the main factor of carotid atherosclerosis. Carotid atherosclerosis and plaque are usually the characteristic manifestations of atherosclerosis. Carotid arteriosclerosis is closely related to stroke, and carotid arteriosclerosis, rupture and detachment of carotid plaques, carotid stenosis and occlusion can all lead to the occurrence of cerebrovascular events. Early detection and evaluation of hyperlipidemia with carotid atherosclerosis by various means can effectively reduce the risk of cardiovascular and cerebrovascular diseases. In order to better serve the vast number of patients, Professor Wang Lei has developed ShenJu granules based on traditional Chinese medicine prescriptions and years of clinical experience. Compared to decoction, ShenJu granules have a higher concentration, are more convenient to carry, and are easy to absorb. They have received unanimous praise from patients in clinical applications.

ELIGIBILITY:
Inclusion Criteria:

1. The patient has informed consent and signed the informed consent form
2. Age between 18-65 years old
3. Meet the diagnostic criteria for hyperlipidemia and accompanied by carotid arteriosclerosis
4. Meet the diagnostic criteria of TCM wet certificate: refer to the scoring standard of TCM Wet Disease Scale

Exclusion Criteria:

1. Severe liver, kidney and cardiac insufficiency
2. Any other serious disease or condition such as: malignant tumor, uncontrolled severe hypertension, diabetic ketoacidosis (acute complication/vascular abnormality), arrhythmia, coagulation abnormalities
3. Have participated in another clinical study within 30 days prior to enrollment or have received a history of randomized ketoacidosis in this study
4. Pregnant women, women preparing to become pregnant and lactating women
5. Patients who are allergic to relevant Chinese medicine ingredients
6. Patients who have had a stent inserted
7. Patients who the investigator determines are not suitable to participate in this study

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-09-20 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Arm and ankle pulse wave velocity | At enrollment versus at day 90
  Measures the degree of carotid artery sclerosis

SECONDARY OUTCOMES:
Blood glucose | At enrollment versus at day 90
  blood glucose in mmol/L
Lipid indexes | At enrollment versus at day 90
  Total cholesterol, triglycerides, low-density lipoprotein, high-density lipoprotein, apolipoprotein (a), free fatty acids
Indicators of carotid atherosclerosis | At enrollment versus at day 90
  IMT value, IMT rate of change, common carotid peak systolic flow rate (PSV), peak diastolic flow rate (EDV), pulsatile index (PI), resistance index (RI)
TCM wet evidence | At enrollment versus at day 90
  Whether it is in the population with phlegm and wetness

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Guangdong Provincial Hospital of Chinese Medicine, Guangzhou, Guangdong
  - WangLei, Guangzhou, Guangdong

IPD SHARING:
Plan to Share IPD: No